CLINICAL TRIAL: NCT06611176
Title: Local Levobupivacaine for Pain Relief After Endoscopic Submucosal Dissection for Esophageal Lesions: a Randomized Controlled Trial
Brief Title: Local LevoBupivacaine for Pain Relief After Endoscopic Submucosal Dissection for Esophageal Lesions
Acronym: BESD-RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laura Boer (Other)
Responsible Party: Sponsor-Investigator, Laura Boer, Principle Investigator, St. Antonius Hospital
Organization: St. Antonius Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-510912-66-00; 2024-510912-66-00 (EU CTIS Number)
Record Dates: First submitted 2024-09-23; First posted 2024-09-24 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-09

CONDITIONS: Endoscopic Submucosal Dissection; Levobupivacaine
Keywords: endoscopic submucosal dissection; ESD; esophagus; analgesic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- No levobupivacaine (No Intervention): ESD without local levobupivacaine
- Levobupivacaine (Experimental): levobupivacaine submucosally injected during esopahgeal esd
  Interventions: Drug: Local levobupivacaine

INTERVENTIONS:
Drug: Local levobupivacaine — submucosal injection of levobupivacaine during esophageal esad
  Arms: Levobupivacaine

SUMMARY:
Endoscopic submucosal dissection (ESD) is commonly performed for (pre)cancerous lesions in the esophagus. Following ESD, post-procedural chest pain is seen in many patients. Studies have shown that local bupivacaine (BP) into the residual submucosal layer of the resection wound after gastric ESD could reduce post-procedural pain rates effectively. Levobupivacaine (LB) is equipotent to BP regarding analgesic effects, but has a better safety profile. No studies have been performed to evaluate the efficacy of LB after esophageal ESD to reduce pain. Therefore, we want to evaluate the effect on post-procedural pain of local application of LB during esophageal ESD.

ELIGIBILITY:
Inclusion Criteria:

* Patients age ≥18 years at time of consent
* Visible lesion in the esophagus, minimum diameter of the lesion ≥20 mm
* Scheduled for esophageal ESD
* Informed consent

Exclusion Criteria:

* Presence of multiple lesions requiring two or more separate endoscopic resections
* History of esophageal surgery other than fundoplications
* History of esophageal ablation therapy
* History of radiotherapy of the esophagus
* Esophageal varices
* Prior endoscopic resection in the same area
* Uncontrolled coagulopathy
* Severe medical comorbidities precluding endoscopy
* Allergy to LB or other amide-type local anaesthesia
* Current regular use of opioids
* Other aetiology causing pain similar to post-ESD pain
* Inability to assess pain due to severe psychiatric or neurological disease
* Insufficient command of Dutch language
* Brugada syndrome
* Incapacitated patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Local levobupivacaine for pain relief after Endoscopic Submucosal Dissection for esophageal lesions: a Randomized Controlled Trial | 90min
  The proportion of patients with major pain within 90 minutes after the procedure comparing the LB and non-LB group. Major pain is defined as a pain score of 4 or higher on a 0-10 Numeric Rating Scale (NRS). The highest pain score reported at any of the three pre-defined time points (30, 60, or 90 minutes after the procedure) will be used to determine if a patient experienced major pain

SECONDARY OUTCOMES:
Local levobupivacaine for pain relief after Endoscopic Submucosal Dissection for esophageal lesions: a Randomized Controlled Trial | 14 days
  Pain scores based on a 0-10 NRS within 90 minutes after the procedure, 6 hours after the procedure and thereafter daily up to day 14.
  * Cumulative pain throughout 14 days based on the area under the curve of a pain versus time plot.
  * Duration of pain, defined as the number of days until pain scores were reported to be 0 on all following days.
  * Daily and overall use of analgesics up to day 14 post-procedurally registered in a patient diary (electronic or on paper).
  * Length of hospital stay in days
  * Incidence of serious adverse events related to LB administration (including allergic reactions to LB).
  * Incidence of adverse events related to LB ad ministration (including allergic reactions to LB).

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - UMCG, Groningen
  - St Antonius Hospital, Nieuwegein
  - UMCU, Utrecht

IPD SHARING:
Plan to Share IPD: Undecided